CLINICAL TRIAL: NCT03231722
Title: The TRIPLETE Study RANDOMIZED PHASE III STUDY OF TRIPLET mFOLFOXIRI PLUS PANITUMUMAB Versus mFOLFOX6 PLUS PANITUMUMAB AS INITIAL THERAPY FOR UNRESECTABLE RAS AND BRAF WILDTYPE METASTATIC COLORECTAL CANCER PATIENTS
Brief Title: First Line mFOLFOXIRI + PANITUMUMAB vs mFOLFOX + PANITUMUMAB IN RAS AND BRAF WT METASTATIC COLORECTAL CANCER PATIENTS
Acronym: TRIPLETE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPLETE
Record Dates: First submitted 2017-07-03; First posted 2017-07-27 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mFOLFOXIRI + Panitumumab; RAS and BRAF wt
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFOX6 + Panitumab (Active Comparator): * Panitumumab 6 mg/kg iv over 60 minutes, day 1 (if the first infusion is tolerated, then subsequent infusions may be administered over 30 to 60 minutes) followed by
  * Oxaliplatin 85 mg/sqm iv over 2 hours, day 1 in two-way with
  * L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 followed by
  * 5-fluorouracil 400 mg/sqm iv bolus, day 1 followed by
  * 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. If no progression occurs, patients will receive maintenance with 5FU/LV plus pan at the same dose used at the last cycle of the induction treatment. 5FU/LV plus pan will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal. The prosecution of pan until disease progression is recommended also if 5-FU is interrupted because of adverse events, patient's refusal or investigator's choice.
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: l-leucovorin; Drug: 5-fluorouracil
- mFOLFOXIRI + Panitumumab (Experimental): * Panitumumab 6 mg/kg iv over 60 minutes, day 1 (if the first infusion is tolerated, then subsequent infusions may be administered over 30 to 60 minutes) followed by
  * Irinotecan 150 mg/sqm iv over 60 minutes day 1, followed by
  * Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with
  * L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 followed by
  * 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. If no progression occurs, patients will receive maintenance with 5FU/LV plus pan at the same dose used at the last cycle of the induction treatment. 5FU/LV plus pan will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal. The prosecution of pan until disease progression is recommended also if 5-FU is interrupted because of adverse events, patient's refusal or investigator's choice.
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: l-leucovorin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Panitumumab — 6 mg/kg iv over 60 minutes, day 1
Drug: Irinotecan — 150 mg/sqm iv over 60 minutes day 1
Drug: Oxaliplatin — 85 mg/sqm iv over 2 hours day 1
  Arms: mFOLFOXIRI + Panitumumab
Drug: l-leucovorin — 200 mg/sqm iv over 2 hours
Drug: 5-fluorouracil — 400 mg/sqm iv bolus, day 1 followed by 2400 mg/sqm 48 h-continuous infusion, starting on day 1;

SUMMARY:
* The association of FOLFOX (5-fluoruracil, folinic acid, and oxaliplatin) and pan is a standard option for the first-line treatment of unresectable RAS and BRAF wt mCRC patients.
* The phase III TRIBE trial recently demonstrated that FOLFOXIRI (5-fluoruracil, folinic acid, oxaliplatin and irinotecan) plus bev significantly prolongs PFS and OS and increases RECIST response rate, ETS and DoR, as compared to FOLFIRI (5-fluoruracil folinic acid, and irinotecan) plus bev. The advantage provided by the intensification of the upfront chemotherapy backbone is independent of RAS and BRAF mutational status.
* Some phase II trials recently assessed the safety and activity of the combination of three-drugs chemotherapy regimens with an anti-EGFR monoclonal antibody. Promising activity results in terms of RECIST response rate and R0 resection rate have been achieved, with some safety concerns with special regards to gastrointestinal toxicity.
* In the phase II randomized MACBETH study the combination of a modified schedule of FOLFOXIRI with cetuximab determined remarkable activity results, with an acceptable and manageable safety profile.
* The optimal duration of the upfront treatment with chemotherapy plus anti-EGFRs is not established. The phase II MACRO-2 trial suggested that interrupting FOLFOX after 4 months while continuing cet alone as maintenance, is a reasonable option.
* Activity parameters (RECIST response rate, ETS, DoR) are clinically relevant endpoints, associated with longer survival, in particular with anti-EGFR moAb-based treatment.

On the basis of these considerations, we designed the present phase III randomized trial of first-line mFOLFOXIRI plus pan versus mFOLFOX6 plus pan in RAS and BRAF wt unresectable mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures and to molecular analyses.
* Histologically proven diagnosis of colorectal cancer.
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* At least one measurable lesion according to RECIST 1.1.
* Availability of a tumour tissue sample (primary tumour and/or metastatic sites).
* Male or female of 18-75 years of age
* ECOG PS ≤2 for patients aged ≤70 years; ECOG PS 0 for patients aged 71 to 75 years.
* Life expectancy of at least 12 weeks
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse.
* RAS (codons 12, 13, 59, 61, 117 and 146 of KRAS and NRAS genes) and BRAF (V600E mutation) wt status of primary colorectal cancer or related metastasis (local or central laboratory assessment).
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥9 g/dl.
* Total bilirubin ≤ 1.5 fold the upper-normal limits (UNL), ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases).
* Creatinine clearance ≥50 mL/min or serum creatinine ≤1.5 x UNL.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception - Contraception, starting with the first dose of study therapy through 180 days after the last dose of treatment.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit
* Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study starting with the first dose of study therapy through 180 days after the last dose of treatment.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

* Will and ability to comply with the protocol.

Exclusion Criteria:

* Previous treatment for metastatic disease.
* Radiotherapy to any site within 4 weeks before the study.
* Previous adjuvant oxaliplatin-containing chemotherapy.
* Previous treatment with EGFR inhibitors.
* Untreated brain metastases or spinal cord compression or primary brain tumours.
* History or evidence upon physical examination of CNS disease unless adequately treated.
* Symptomatic peripheral neuropathy > 1 grade NCIC-CTG criteria.
* Creatinine clearance < 50 mL/min or serum creatinine >1.5 x UNL.
* Clinical signs of malnutrition.
* Neutrophils <1.5 x 109/L, Platelets <100 x 109/L, Hgb <9 g/dl.
* Diagnosis of interstitial pneumonitis or pulmonary fibrosis.
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration.
* Clinically significant (e.g. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication.
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness, or hepatitis B or C.
* Definite contraindications for the use of corticosteroids and antihistamines as premedication.
* History of severe allergic reactions or hypersensitivity to trial drugs or any of their excipients.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 180 days after the last trial treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 12 months
  the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Toxicity Rate | 24 months
  the percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 4.0)
Toxicity Rate | 24 months
  the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 4.0)
Progression Free Survival | 24 months
  the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. Documentation of disease progressive disease is defined as per RECIST 1.1 criteria based on investigator assessment
Overall Survival | 48 months
  the time from randomization to the date of death due to any cause
Centrally assessed Overall response rate | 12 months
  the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria based on central re-evaluation of CT scan images.
Early Tumour Shrinkage Rate | up to 2 months from randomization
  the percentage of patients, relative to the total of the enrolled subjects, achieving a ≥20% decrease in the sum of diameters of RECIST target lesions at week 8 compared to baseline.
Deepness of Response | 12 months
  the relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline.
R0 Resection Rate | 12 months
  the percentage of patients, relative to the total of enrolled subjects, undergoing secondary R0 resection of metastases

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Cremolini, MD, PhD, Study Chair — U.O. Oncologia Medica 2 Universitaria - Azienda Ospedaliero-Universitaria Pisana Dipartimento di Ricerca Traslazionale e Nuove Tecnologie - Università di Pisa Istituto Toscano Tumori
Locations (4):
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Fondazione IRCCS Istituto Oncologico Veneto, Padua
  - A.O. Universitaria Pisana - Pisa (Pi) Oncologia Medica, Pisa
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conca V, Rossini D, Antoniotti C, Lonardi S, Pietrantonio F, Moretto R, Antonuzzo L, Randon G, Lavacchi D, Pozzo C, Marmorino F, Bergamo F, Tamburini E, Passardi A, Fazio R, Murgioni S, Borelli B, Buonadonna A, Germani MM, Formica V, Carullo M, Bordonaro R, Aprile G, Zaniboni A, Masi G, Boni L, Cremolini C. Upfront Modified FOLFOXIRI Plus Panitumumab for RAS/BRAF Wild-Type Metastatic Colorectal Cancer: Final Results of the Phase III TRIPLETE Study. J Clin Oncol. 2026 Feb 10;44(5):361-369. doi: 10.1200/JCO-25-01337. Epub 2026 Jan 8. PMID 41505697
- [Derived] Sposito C, Pietrantonio F, Maspero M, Di Benedetto F, Vivarelli M, Tisone G, De Carlis L, Romagnoli R, Gruttadauria S, Colledan M, Agnes S, Ettorre G, Baccarani U, Torzilli G, Di Sandro S, Pinelli D, Caccamo L, Sartore Bianchi A, Spreafico C, Torri V, Mazzaferro V. Improving Outcome of Selected Patients With Non-Resectable Hepatic Metastases From Colorectal Cancer With Liver Transplantation: A Prospective Parallel Trial (COLT trial). Clin Colorectal Cancer. 2023 Jun;22(2):250-255. doi: 10.1016/j.clcc.2023.01.003. Epub 2023 Feb 3. PMID 36822922
- [Derived] Rossini D, Antoniotti C, Lonardi S, Pietrantonio F, Moretto R, Antonuzzo L, Boccaccino A, Morano F, Brugia M, Pozzo C, Marmorino F, Bergamo F, Tamburini E, Passardi A, Randon G, Murgioni S, Borelli B, Buonadonna A, Giordano M, Fontanini G, Conca V, Formica V, Aglietta M, Bordonaro R, Aprile G, Masi G, Boni L, Cremolini C. Upfront Modified Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan Plus Panitumumab Versus Fluorouracil, Leucovorin, and Oxaliplatin Plus Panitumumab for Patients With RAS/BRAF Wild-Type Metastatic Colorectal Cancer: The Phase III TRIPLETE Study by GONO. J Clin Oncol. 2022 Sep 1;40(25):2878-2888. doi: 10.1200/JCO.22.00839. Epub 2022 Jun 6. PMID 35666229
- [Derived] Borelli B, Moretto R, Lonardi S, Bonetti A, Antoniotti C, Pietrantonio F, Masi G, Burgio V, Marmorino F, Salvatore L, Rossini D, Zaniboni A, Zucchelli G, Martignetti A, Di Battista M, Pella N, Passardi A, Boccaccino A, Leone F, Colombo C, Granetto C, Vannini F, Marsico VA, Martinelli E, Antonuzzo L, Vitello S, Delliponti L, Boni L, Cremolini C, Falcone A. TRIPLETE: a randomised phase III study of modified FOLFOXIRI plus panitumumab versus mFOLFOX6 plus panitumumab as initial therapy for patients with unresectable RAS and BRAF wild-type metastatic colorectal cancer. ESMO Open. 2018 Jul 9;3(4):e000403. doi: 10.1136/esmoopen-2018-000403. eCollection 2018. PMID 30018814